CLINICAL TRIAL: NCT04180033
Title: Diagnostic Yield of Colonoscopy Surveillance in Testicular Cancer Survivors Treated With Platinum-based Chemotherapy
Acronym: CATCHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M19CTR
Record Dates: First submitted 2019-11-06; First posted 2019-11-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2020-02

CONDITIONS: Testicular Cancer; Colorectal Neoplasms
Keywords: Colonoscopy surveillance
MeSH Terms: conditions — Testicular Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be invited to undergo a colonoscopy surveillance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colonoscopy surveillance in TC survivors (Other): TC survivors treated with platinum-based chemotherapy will be invited to undergo a colonoscopy surveillance.
  Interventions: Diagnostic Test: Colonoscopy surveillance

INTERVENTIONS:
Diagnostic Test: Colonoscopy surveillance — Participants will be asked to undergo a first colonoscopy surveillance.
  Other Names: Fecal immunochemical test (FIT)

SUMMARY:
Testicular cancer (TC) survivors treated with platinum-based chemotherapy have an increased risk of colorectal cancer (CRC) (hazard ratio (HR) 3.9 for platinum-containing chemotherapy versus no platinum-containing chemotherapy, 95% confidence interval 1.7-8.9). Colonoscopy screening can reduce CRC incidence and mortality. Given this increased risk of CRC, colonoscopy surveillance should be considered for TC survivors treated with platinum-based chemotherapy.

The aim of this study is to evaluate the diagnostic yield of advanced colorectal neoplasia during colonoscopy surveillance in TC survivors treated with platinum-based chemotherapy. The secondary objectives are to determine cost-effectiveness and burden of colonoscopy. Furthermore, the molecular profile of advanced neoplasia will be evaluated to create insight into the carcinogenesis. The effectiveness of fecal immunochemical testing (FIT) will be evaluated with colonoscopy as a reference. Finally, blood plasma platinum-levels will be determined to examine a potential correlation with the outcome of the ccolonoscopy.

DETAILED DESCRIPTION:
Rationale: Testicular cancer (TC) survivors have an increased risk of various second primary malignancies. A recent cohort study showed that platinum-based chemotherapy was associated with increased risk of colorectal cancer (CRC) in a dose dependent manner (hazard ratio (HR) 3.9 for platinum-containing chemotherapy versus no platinum-containing chemotherapy, 95% confidence interval 1.7-8.9). Colonoscopy screening can reduce CRC incidence and mortality. Given this increased risk of CRC, colonoscopy surveillance should be considered for TC survivors treated with platinum-based chemotherapy. However, the diagnostic yield, cost-effectiveness and burden of colonoscopy in TC survivors treated with platinum-based chemotherapy has never been assessed. Additionally, the molecular profile of advanced neoplastic lesions and CRC in TC survivors treated with platinum-based chemotherapy has not been established but can provide valuable insight into CRC carcinogenesis in this group of patients. Also the effectiveness of fecal tests has not been evaluated among TC survivors treated with platinum-based chemotherapy compared to that among population controls.

Objective: The primary objective of this study is to assess the diagnostic yield of colonoscopy surveillance in TC survivors treated with platinum-based chemotherapy. The secondary objectives are 1) to evaluate the molecular characteristics of colorectal (advanced) neoplasia in TC patients in relation to the cumulative doses of/ level of plasma cisplatin, in order to improve the understanding of CRC carcinogenesis following cisplatin exposure, 2) to determine the association of platinum levels in plasma with cumulative administered cisplatin doses as well as with presence of colorectal (advanced) neoplasia at colonoscopy and to determine the platinum amount in the colorectal tissue derived during primary colonoscopy screening, 3) to evaluate the cost-effectiveness and burden of colonoscopy. Our 4th secondary objective is to assess the effectiveness of a stool test for CRC screening in TC survivors compared to standard colonoscopy.

Study design: A multicentre prospective cross-sectional screening study.

Study population: TC survivors will be derived from an established, well-defined multicentre cohort. Inclusion criteria of this study are 1) participants should have been treated for TC in a participating Dutch hospital before the age of 50 years, 2) treatment consisted of at least three cycles of platinum-based chemotherapy (cisplatin) with or without additional radiotherapy, 3) participants should be at least 8 years after start of treatment, with a minimum age at first colonoscopy screening of 35 years, 4) the maximum age at participation is 75 years, 5) detection and potential treatment of advanced colorectal neoplasia is considered beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TC before age of 50 years
* Treatment of primary TC consisting at least: three cycles of platinum-based chemotherapy consisting of cisplatin
* At least 8 years after initial treatment
* At least 35 years of age and not older than 70 75 years
* Detection and potential treatment of advanced colorectal neoplasia is considered beneficial

Exclusion Criteria:

* A history of a proctocolectomy
* Colonoscopy surveillance for other indications (including hereditary CRC syndrome, familial CRC syndrome, inflammatory bowel disease, history of colorectal adenoma or CRC). Result of the prior colonoscopy will be put in the database and used for additional analyses
* Having received a colonoscopy in the past three years
* Currently receiving cytotoxic treatment or radiotherapy for malignant disease
* Coagulopathy (prothrombin time <50% of control; partial tromboplastin time >50 seconds) or anticoagulants (fenprocoumon, acenocoumarol, platelet aggregation inhibitors or new oral anticoagulants) that cannot be stopped or safely bridged if necessary
* Comorbidity leading to an impaired physical performance (World health organization (WHO) performance status 3-4) or mental retardation
* Limited Dutch language skills
* No informed consent

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield advanced colorectal neoplasia | 2 years
  Diagnostic yield of advanced colorectal neoplasia detection by a first colonoscopy surveillance.

SECONDARY OUTCOMES:
Features of colorectal neoplasia as classified during colonoscopy | 2 years
  Colorectal neoplasia characteristics including endoscopic features (morphology, prevalence, size and location)
Molecular features of colorectal neoplasia and normal mucosa as evaluated histopathologically, molecular and by immunohistochemistry | 6 months
  The molecular profile of advanced colorectal neoplasia and normal colorectal tissue will be evaluated by immunohistochemistry and molecular pathology
Platinum levels in plasma | 2 years
  Measure platinum in plasma and possibly in FFPE material of CRC
Fecal immunochemical test (FIT) | 2 years
  Performance (sensitivity/specificity/positive predictive value/negative predictive value) of the fecal immunochemical test (FIT) stool test to detect advanced colorectal neoplasia will be evaluated using the colonoscopy as reference standard.
Determination of the most cost-effectiveness strategy for colonoscopy surveillance by using the MISCAN model | 3 months
  Cost-effectiveness analysis of colonoscopy screening using the microsimulation screening analysis (MISCAN) model to evaluate the most cost-effective strategy.
Quality of life of participant before and after colonoscopy | 2 years
  Quality of life before and after colonoscopy will be evaluated by validated questionnaires (EQ-5D). This is a standardized instrument to evaluate five health categories (mobility, self care, daily activities, pain/discomfort and fear/depression). The items can be scored in three values; no/some/a lot of problems. A higher score represents a worse outcome.
  Furthermore, the health will be scored on a 0 to 100 scale. A higher score will correspond with a better health interpreted health of the participant.
Worries about cancer | 2 years
  The cancer worry scale will be used to evaluate the worries about cancer (4 point scale; 1 (hardly never) to 4 (regularly() via a questionnaire before colonoscopy
Burden of colonoscopy | 2 years
  Two questionnaire (before and after colonoscopy) will be performed to evaluate the expected and experienced burden of colonoscopy using a 5-point scale (1 - Hardly to 5 - Very)

CONTACTS AND LOCATIONS:
Overall Officials: Monique van Leerdam, MD PhD, Principal Investigator — Antoni van Leeuwenhoek Hospital
Locations (4):
- Netherlands (4):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Breekveldt ECH, Ykema BLM, Huitema ADR, Gietema JA, Beijnen JH, Snaebjornsson P, Schaapveld M, van Leeuwen FE, Rosing H, van Leerdam ME; CATCHER study working group. Platinum retention in plasma, urine, and normal colonic mucosa in cisplatin-treated testicular cancer survivors. PLoS One. 2024 Nov 14;19(11):e0312994. doi: 10.1371/journal.pone.0312994. eCollection 2024. PMID 39541403
- [Derived] Ykema BLM, Bisseling TM, Spaander MCW, Moons LMG, van der Biessen-van Beek D, Saveur L, Kerst M, Mulder SF, de Wit R, Zweers D, Meijer GA, Beijnen JH, Lansdorp-Vogelaar I, van Leeuwen FE, Snaebjornsson P, van Leerdam ME. Diagnostic yield of colonoscopy surveillance in testicular cancer survivors treated with platinum-based chemotherapy: study protocol of a prospective cross-sectional cohort study. BMC Gastroenterol. 2021 Feb 12;21(1):67. doi: 10.1186/s12876-021-01639-2. PMID 33579196